CLINICAL TRIAL: NCT07140237
Title: The Influence and Regulatory Role of Exogenous and Endogenous Oxytocin on Top-down Attention in Humans
Brief Title: The Effect of Oral Oxytocin and Atosiban on Top-down Attention ( OTAtosiban )
Acronym: OTAtosiban
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN99
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adult Male
Keywords: Oxytocin; Atosiban; Eye-tracking; Autistic trait; Oxytocin; Atosiban; Eye-tracking; Autistic trait; attention
MeSH Terms: interventions — atosiban

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design experiment including 5 treatment groups receiving oral oxytocin, atosiban, or placebo interventions prior to performing antisaccade task.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Oxtocin 24IU group (Experimental): Interventions are placebo followed after 15 minutes by the lower does (24IU) oxytocin
  Interventions: Drug: Oxytocin lower does (24IU); Drug: Placebo
- atosiban group (Experimental): Interventions are placebo followed after 15 minutes by 150ug atosiban
  Interventions: Drug: Atosiban; Drug: Placebo
- placebo group (Placebo Comparator): Interventions are placebo followed after 15 minutes by another placebo
  Interventions: Drug: Placebo
- Oxytocin 48IU group (Experimental): Interventions are placebo followed after 15 minutes by the higher 48IU oxytocin does
  Interventions: Drug: Oxytocin higher does (48IU); Drug: Placebo
- Atosiban and 24IU oxytocin group (Experimental): Interventions are atosiban 150ug followed after 15 minutes by the lower (24IU) does of oxytocin
  Interventions: Drug: Oxytocin lower does (24IU); Drug: Atosiban

INTERVENTIONS:
Drug: Oxytocin lower does (24IU) — Oxytocin (24IU) will be administered as a lingual spray (6, 0.1puffs (4IU per puff) of spray on and under the tongue)
  Arms: Atosiban and 24IU oxytocin group; Oxtocin 24IU group
Drug: Oxytocin higher does (48IU) — Oxytocin (48IU) will be administered as a lingual spray (6, 0.1ml sprays (8IU per puff) on and under the tongue)
  Arms: Oxytocin 48IU group
Drug: Atosiban — 150ug atosiban administered by lingual sprays (6, 0.1ml sprays on and under the tongue)
  Arms: Atosiban and 24IU oxytocin group; atosiban group
Drug: Placebo — Placebo administered as a lingual spray (6, 0.1puffs (4IU per puff) of spray on and under the tongue). Placebo has the same composition of 0.9% saline and glycerol as for oxytocin and the atosiban interventions.
  Arms: Oxtocin 24IU group; Oxytocin 48IU group; atosiban group; placebo group

SUMMARY:
The main aim of the present study is to investigate whether orally (lingual spray) administered oxytocin influences human top-down attention via oxytocin receptors and whether its effects are dose- and task-dependent.

DETAILED DESCRIPTION:
In a placebo-controlled double-blind between-subject design experiment, investigators plan to investigate whether oral (lingual spray) oxytocin influences human top-down attention via the oxytocin receptor and whether its effects are dose- and task-dependent. Subjects complete questionnaires in Chinese versions before treatment administration, including Behavioral Activation System scale, Behavioral Inhibition System scale,Trait Anxiety Inventory, State Anxiety Inventory, Liebowitz Social Anxiety Scale, Beck Depression Inventory, Autism Spectrum Quotient. Then the first blood (6ml via indwelling medial cubital vein catheter) and saliva (1-2 ml, passive drool) samples are collected, followed by the first self-administered medication (three sublingual and three supragingival administrations, alternating separated by 30 seconds). After a 15-minute interval, the second medication is administered, with a second blood sample collected immediately afterwards. Subjects then remain in the lab for 30 minutes (mobile phone use and conversation with experimenters are prohibited during this period). Behavioral experiment (antisaccade) commences after the third blood collection. During these phases, subjects' latency of correct trials, error rate and pupil size in response to stimuli will be measured using eye tracking equipment. Immediately after completion of the paradigm subjects will complete the state anxiety questionnaire again to assess treatment/paradigm effects on anxiety.

A Mixed linear model, followed by appropriate post-hoc analyses will be used on eye-tracking and other data to assess treatment effects. Correlation analysis will be used to assess associations between latency of correct trials in prosaccade and error rate in antisaccade in the different groups. Investigators make the following hypotheses according to our previous studies: first, oral oxytocin treatment will dose-dependently decrease top-down attention to social but also non-social stimuli; secondly, oxytocin concentrations will be dependent on the dose of oral administration and will not be influenced by oral administration of the oxytocin receptor antagonist (atosiban) administration; thirdly, atosiban is anticipated to have the opposite effect of oral oxytocin and may not interfere with top-down attention; fourthly, oxytocin treatment will increase pupil diameter while viewing social stimuli; fifthly, there will be treatment- dependent effects on post-task state anxiety scores; lastly, antisaccade performance in each group might be influenced by subjects' scores on autistic traits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* History of or current neurological/psychiatric disorders;
* Use of psychotropic medications (including nicotine)
* Visual impairments

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects without past or current psychiatric or neurological disorders
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Error rates in prosaccade and antisaccade trials | Starting 45 minutes post-treatment subjects will complete the eye-tracking task with data on numbers of prosaccade and antisaccade errors being collected continuously over a period of 35 minutes.
  Error rates in prosaccade and antisaccade using eye- tracking technique
Responses latencies for prosaccades and antisaccades | Starting 45 minutes post-treatment subjects will complete the eye-tracking task with data on prosaccade and antisaccade response times taken continuously during the 35 minute task
  response latencies for correct first saccades will be measured on each prosaccade or antisaccade trial using eye-tracking

SECONDARY OUTCOMES:
Oxytocin concentration | On the day of the experiment blood and saliva samples will be taken at time 0 (baseline) immediately prior to the first treatment, a 2nd sample will be taken at 15 minutes and a 3rd sample at 45 minutes post-treatment.
  OT concentrations will be measured in blood (plasma) samples (6ml) taken from indwelling catheter in median cubital vein and saliva samples (1-2ml) taken using passive drool. OT concentrations will be measured using appropriate essays.
Pupil size | Starting 45 minutes post-treatment continuous eye-tracking will be used to measure changes in pupil size during the whole of the 35 minute antisaccade task
  Pupil size will be measured during antisaccade task using eye-tracker
State anxiety | On the day of the experiment subjects will complete the questionnaire immediately prior to treatment at time 0 (baseline) and again 75 minutes post-treatment after completion of the antisaccade task
  State anxiety will be measured using a questionnaire (40 self-report question-state-trait-anxiety inventory, with total scores ranging from 20-80, where higher scores indicate greater anxiety).
Correlation between prosaccade latency and antisaccade errors | Starting 45 minutes post-treatment subjects will complete the eye-tracking task with data being collected continuously over a 35 minute period
  The correlation between two of the primary outcome measures (prosaccade latencies and antisaccade errors) taken during trials will be analyzed using the Spearman correlation test for each treatment group. Differences between correlations in the groups will be assessed using Fisher's z tests

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared with other qualified researchers upon request